CLINICAL TRIAL: NCT02489799
Title: Utilizing Advance Care Planning Videos to Empower Perioperative Cancer Patients and Families
Acronym: ACPvideo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: J1549; IRB00047112 (Other: JHMIRB)
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Cancer
Keywords: advance care planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Advance care planning video
  Interventions: Behavioral: Advance care planning video
- Control (Placebo Comparator): Control video - no advance care planning content
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Advance care planning video — This is a video involving interviews with patients, a family member, two surgeons, an anesthesiologist, and an ICU nurse; these interviewees describe the typical events during a hospitalization for a major surgery and encourage the viewer to do some planning before surgery - the planning includes: (i) naming a person to make decisions for the participant, (ii) having a conversation with that person about goals and values, and (iii) continuing that conversation with the participant's surgeon.
  Arms: Intervention
Behavioral: Control video — This is a video showing the history of The Johns Hopkins Hospital and emphasizing that The Johns Hopkins Hospital is a great place to receive medical care.
  Arms: Control

SUMMARY:
Through close engagement with our patient and family member co-investigators, the investigators have developed a video-based advance care planning aid for cancer patients and their family members who are preparing for major surgery. In this study, patients are randomized to see either the intervention video (involving advance care planning-related content) or a control video (no advance care planning-related content) prior to surgery. The investigators hypothesize that the video will lead to more and better preoperative discussions between the patient and surgeon that are related to advance care planning. The investigators also hypothesize that seeing the advance care planning-related video will decrease perioperative anxiety and depression scores.

DETAILED DESCRIPTION:
Many cancer patients pursue aggressive surgery in the hope of cancer cure or life prolongation. However, in doing so, patients and families may avoid advance care planning; they do not discuss specific goals and wishes should disease progress despite surgery. Moreover, a subset of patients become critically ill following surgery, and family members must make life-and-death decisions without knowing patient wishes. Preoperative advance care planning-facilitating patient and family discussions concerning perioperative goals, hopes, and fears-could empower patients and families to better choose which therapies and procedures they want outside of the initial surgery and for the months following surgery. Advance care planning aids exist, but none were developed for or evaluated in a surgical patient population. Furthermore, video-based advance care planning tools are an innovative way to better empower patients and families. Previous research shows that, with the aid of an advance care planning video, patients and families are more knowledgeable about treatment options and more comfortable with making decisions. Moreover, when better educated, these patients and families frequently choose less aggressive therapies.

However, video-based advance care planning tools have not been developed or tested in a surgical patient population. The investigators have developed and now will evaluate a video-based advance care planning aid for cancer patients and families pursing aggressive surgical cancer treatment. The investigators hypothesize that, in patients and family members, the video-based decision aid will facilitate better preoperative discussions about advance care planning between the patient and surgeon and decrease anxiety and depression after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older of study surgeons who are scheduled to have a surgical procedure identified by study surgeons to the study team.
* Patients willing to give informed consent, ability to speak English, reasonably able to read a newspaper or book (without sight impairment); reasonable able to listen to radio, television (without hearing impairment).

Exclusion Criteria:

* Age <18 years old, non-English speaking patients who are not identified by participating surgeons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Aslakson, MD PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Through mandated reporting by the Patient-Centered Outcomes Research Institute (PCORI), our data will be shared via their website.

REFERENCES:
- [Derived] Aslakson RA, Isenberg SR, Crossnohere NL, Conca-Cheng AM, Moore M, Bhamidipati A, Mora S, Miller J, Singh S, Swoboda SM, Pawlik TM, Weiss M, Volandes A, Smith TJ, Bridges JFP, Roter DL. Integrating Advance Care Planning Videos into Surgical Oncologic Care: A Randomized Clinical Trial. J Palliat Med. 2019 Jul;22(7):764-772. doi: 10.1089/jpm.2018.0209. Epub 2019 Apr 9. PMID 30964385
- [Derived] Isenberg SR, Crossnohere NL, Patel MI, Conca-Cheng A, Bridges JFP, Swoboda SM, Smith TJ, Pawlik TM, Weiss M, Volandes AE, Schuster A, Miller JA, Pastorini C, Roter DL, Aslakson RA. An advance care plan decision support video before major surgery: a patient- and family-centred approach. BMJ Support Palliat Care. 2018 Jun;8(2):229-236. doi: 10.1136/bmjspcare-2017-001449. Epub 2018 Mar 18. PMID 29555812
- [Derived] Aslakson RA, Isenberg SR, Crossnohere NL, Conca-Cheng AM, Yang T, Weiss M, Volandes AE, Bridges JFP, Roter DL. Utilising advance care planning videos to empower perioperative cancer patients and families: a study protocol of a randomised controlled trial. BMJ Open. 2017 Jun 6;7(5):e016257. doi: 10.1136/bmjopen-2017-016257. PMID 28592584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 45 | 47
Presurgical Consent Visit (V2) | 40 | 39
Postsurgical One Week Visit (V3) | 40 | 39
Completed | 36 | 38
Not Completed | 9 | 9
Not completed — Lost to Follow-up | 4 | 1
Not completed — Failure to Maintain Eligibility | 4 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (13.0) | 59.5 (12.4) | 60.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 43 | 46 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 38 | 41 | 79
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Primary Diagnosis [Count of Participants; unit: Participants]
  Pancreatic Cancer | 15 | 14 | 29
  Colon Cancer | 5 | 3 | 8
  Hepatobiliary and other Gastrointestinal Cancer | 9 | 16 | 25
  Gynecological Cancers | 6 | 6 | 12
  Sarcoma | 7 | 6 | 13
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Measured ACP Content in the Presurgical Consent Visit
Description: The RIAS scoring system using an audio-recording of a conversation to evaluate conversation content.
Time Frame: Approximately one week after study enrollment.
Population: Of note, the sample size is smaller for this outcome as our study did not collect recordings for all participants enrolled at the baseline visit. The reasons we did not collect the recordings include scheduling of emergent surgery without time to record, human and technology error, and patient preference.
Measure: Count of Units; unit: Recordings
Units Other Than Participants: Recordings
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
Number analyzed (Recordings) | 30 | 31
Recordings
  Death (Long-Term) | 6 | 5
  Goals | 10 | 8
  Video | 2 | 1
  Alternate Medical Decision Maker | 7 | 3

2. Primary Outcome: Measured Patient Centeredness in the Presurgical Consent Visit
Description: The RIAS scoring system using an audio-recording of a conversation to evaluate the nature of the conversation between surgeon and patient. The patient-centeredness summary score is a ratio of statements that reflect the psychosocial and socio-emotional elements of exchange about the lived illness experience of patients relative to statements that reflect a more biomedical and disease focused perspective. This score reflects the encounter as a whole, rather than an individual's dialogue. A value greater than one indicates a more patient-centered encounter; whereas, a value less than one indicates a more biomedical encounter.
Time Frame: Approximately one week after study enrollment.
Population: Audio recordings of a presurgical consent visit conversation between a surgeon and patient.
Measure: Mean (Standard Deviation); unit: Patient Centeredness Score
Units Other Than Participants: Audio Recordings
Arm/Group | Intervention | Control
Number analyzed (Participants) | 30 | 31
Number analyzed (Audio Recordings) | 30 | 31
Patient Centeredness Score | 0.70 (0.34) | 0.69 (0.28)
Statistical Analysis 1: Comparison: Intervention vs Control; We employed two ways of interpreting this data. The first treats the outcome continuously, which is described in the results section. Here we describe the outcome treating it as a ratio. We created a variable representing the numerator of the ratio (type 1) and the denominator of the ratio (type 2) thereby treating the information in both the numerator and denominator as random (each a Poisson variable); Test type: Equivalence — The study was powered based on two former studies utilizing RIAS, (both powered =.8 and alpha =.05). With a 0.6 effect size, the required sample size is 72 patients (36 per group) for a one-tailed test of study hypotheses (power =.8 and alpha =.05); p = 0.545, Poisson model using GEE; We fit a Poisson model using generalized estimating equations. No adjustments were made for degrees of freedom; Incidence Rate Ratio = 1.06, 95% CI 2-sided [0.87 to 1.30] — The incidence rate ratio compares intervention to control

3. Secondary Outcome: Hospital Anxiety and Depression Scores Across Study Arms Throughout the Study Period
Description: This validated metric consists of two sub scales: one for symptoms of anxiety, and the other for symptoms of depression. Each subscale, consisting of seven questions, results in a score ranging from 0, indicating no distress, to 21, indicating maximum distress; a score higher than 7 indicates clinically meaningful anxiety or depression. Overall HADS scores, encompassing both subscales, results in a total score of 0 (no mood symptoms ) to 42 (maximal mood symptoms).
Time Frame: Enrollment, one week after enrollment, one week after surgery, one month after surgery
Population: At each milestone of data collection, a number of participants were unable to complete the HADS questionnaire due to one of a number of factors including complicated medical course, attrition, or loss of eligibility.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 47
units on a scale
  Baseline Visit (V1) | 9.4 (5.1) | 9.9 (5.7)
  Presurgical Consent Visit (V2): number analyzed (Participants) | 34 | 31
  Presurgical Consent Visit (V2) | 9.4 (7.0) | 9.3 (5.5)
  Postsurgical One Week Visit (V3): number analyzed (Participants) | 37 | 37
  Postsurgical One Week Visit (V3) | 11.5 (6.8) | 13.0 (8.2)
  Postsurgical One Month Visit (V4): number analyzed (Participants) | 36 | 37
  Postsurgical One Month Visit (V4) | 9.6 (7.1) | 10.9 (6.7)

4. Secondary Outcome: Iowa Goals of Care Across Study Arms Throughout the Study Period
Description: This metric enables respondents to verify why they are seeking medical care. The most selected goal at all visits was "Cure my medical condition." We have reported the number of participants in each group who selected this goal at each time point.
Time Frame: Enrollment, one week after enrollment, one week after surgery, one month after surgery
Population: At each milestone of data collection, a number of participants were unable to complete the Iowa Goals of Care questionnaire due to one of a number of factors including complicated medical course, attrition, or loss of eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 47
Participants
  Baseline Visit (V1) | 43 | 46
  Presurgical Consent Visit (V2): number analyzed (Participants) | 34 | 31
  Presurgical Consent Visit (V2) | 33 | 29
  Postsurgical One Week Visit (V3): number analyzed (Participants) | 38 | 37
  Postsurgical One Week Visit (V3) | 34 | 34
  Postsurgical One Month Visit (V4): number analyzed (Participants) | 36 | 37
  Postsurgical One Month Visit (V4) | 34 | 35

5. Secondary Outcome: Helpfulness of the Video Across Study Arms
Description: This Likert scale evaluates respondent beliefs about the helpfulness of the video.
Time Frame: One week after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 31
Participants
  Very Helpful | 14 | 12
  Somewhat Helpful | 14 | 9
  A Little Helpful | 6 | 2
  Not Helpful | 0 | 8

6. Secondary Outcome: Comfort With the Video Across Study Arms
Description: This Likert scale evaluates respondent beliefs about their comfort in viewing the video.
Time Frame: One week after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 31
Participants
  Very Comfortable | 25 | 22
  Somewhat Comfortable | 7 | 8
  Somewhat Uncomfortable | 2 | 1
  Very Uncomfortable | 0 | 0

7. Secondary Outcome: Recommendation of the Video to Others Across Study Arms
Description: This Likert scale evaluates respondent beliefs about whether they would recommend the video to others.
Time Frame: One week after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 31
Participants
  Definitely Recommend | 21 | 16
  Probably Recommend | 11 | 10
  Probably Would Not Recommend | 2 | 4
  Definitely Would Not Recommend | 0 | 1

8. Secondary Outcome: Patient and Provider Satisfaction Scores Across Study Arms
Description: The satisfaction score, as the sum of the scores of six questions (all in Likert scale), ranges from 6 to 30, with a higher score indicating higher level of satisfaction.
Time Frame: One week after enrollment
Population: In two instances, the surgeon was unable to complete the satisfaction scale. This explains why there are fewer surgeon perceptions reported than patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 31
units on a scale
  Patient Self-Reported Satisfaction | 27.2 (5.6) | 27.8 (4.5)
  Surgeon Self-Reported Satisfaction: number analyzed (Participants) | 32 | 31
  Surgeon Self-Reported Satisfaction | 24.9 (2.9) | 24.1 (4.7)

9. Secondary Outcome: Prevalence of Participants Who Acknowledge Having Named a Surrogate Decision Maker Across Study Arms Throughout the Study Period
Description: This tracks which participants report having named a surrogate decision maker
Time Frame: Enrollment, one month after surgery
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 47
Participants
  Baseline Visit (V1): Have Not Identified a Medical Decision Maker | 9 | 11
  Baseline Visit (V1): Have Identified a Medical Decision Maker | 36 | 36
  Postsurgical One Month Visit (V4): number analyzed (Participants) | 36 | 38
  Postsurgical One Month Visit (V4): Have Not Identified a Medical Decision Maker | 2 | 0
  Postsurgical One Month Visit (V4): Have Identified a Medical Decision Maker | 34 | 38

10. Secondary Outcome: Prevalence of Participants Who Acknowledge Having a Conversation With Their Surrogate Decision Maker Regarding Advance Care Planning Across Study Arms Throughout the Study Period
Description: This tracks which participants report having had an advance care planning-related conversation with their surrogate decision maker.
Time Frame: Enrollment, one month after surgery
Population: This question was only asked to participants who reported having designated a medical decision maker.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 45 | 47
Participants
  Baseline Visit (V1): number analyzed (Participants) | 36 | 36
  Baseline Visit (V1): No | 6 | 7
  Baseline Visit (V1): Yes, over 6 months ago | 4 | 6
  Baseline Visit (V1): Yes, within the last 6 months | 26 | 23
  Postsurgical One Month Visit (V4): number analyzed (Participants) | 34 | 38
  Postsurgical One Month Visit (V4): No | 2 | 3
  Postsurgical One Month Visit (V4): Yes, over 6 months ago | 0 | 5
  Postsurgical One Month Visit (V4): Yes, within the last 6 months | 32 | 30

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47
Other Adverse Events (participants affected / at risk) | 0/45 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No